CLINICAL TRIAL: NCT04926779
Title: Open Label, Single-Center Study Utilizing BIOZEK COVID-19 Antigen Rapid Test: Comparison of Biozek COVID-19 Antigen Rapid Test Results Performed on Self-collected Samples by the Subjects, to Results of COVID-19 RT-PCR as a Standard of Care
Brief Title: Study Utilizing BIOZEK COVID-19 Antigen Rapid Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mach-E B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Biozek-ARTC-US/002/4-12-2021
Record Dates: First submitted 2021-06-11; First posted 2021-06-15 (Actual); Results first posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Covid-19 Testing
Keywords: Covid-19; Antigen; Rapid; Test
MeSH Terms: conditions — COVID-19; Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: Biozek Covid-19 Antigen Rapid Test (Saliva) — Self-collection of nasopharyngeal and saliva samples and self test performance - Biozek Covid-19 Antigen Rapid Test (Saliva) and Biozek Covid-19 Antigen Rapid Test (Nasopharyngeal Swab). Both procedures are supervised by trained study personnel.
  Other Names: Biozek Covid-19 Antigen Rapid Test (Nasopharyngeal Swab)

SUMMARY:
This is a research study to evaluate the Sensitivity and Specificity of BIOZEK COVID-19 Antigen Rapid Test (Saliva) and BIOZEK COVID-19 Antigen Rapid Test (Nasopharyngeal Swab) on samples that are self-collected; and to perform analysis to compare results. In addition, to obtain RT-PCR test results, performed prior to enrollment, and compare all three results.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be ≥18 years of age and have had an RT-PCR test performed prior to enrollment.
* Subjects must be able to understand and willingly sign a written informed consent. Additionally, participants need to meet at least 1 of the criteria listed below:

  * Currently experiencing symptoms of COVID-19.
  * Be clinically diagnosed or suspected to have COVID-19.
  * Recent past (3 weeks) exhibited symptoms of COVID-19.
  * Be capable of performing a self-collection of a nasopharyngeal sample with use of nasal swab kit.
  * Be capable of performing a self-collection of an oral fluid sample with use of oral fluid collection kit.
  * Interacted with a COVID-19 positive individual.

Exclusion Criteria:

Subjects who meet any of the following exclusion criteria may not be enrolled in this study:

* Cannot perform self-collection of a nasopharyngeal sample with use of nasal swab kit.
* Cannot perform self-collection of an oral fluid sample with use of oral fluid collection kit.
* Have a deviated nasal septum.
* Cognitively impaired individuals resulting in the inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2022-11-04 (Actual); Study Completion 2022-11-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Mobile Covid Services LLC, Flushing, New York
  - Quality Research and Invention LLC, Southampton, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- BIOZEK COVID-19 Antigen Rapid Test: BIOZEK COVID-19 Antigen Rapid Test (Saliva) and BIOZEK COVID-19 Antigen Rapid Test (Nasopharyngeal Swab) was performed by subjects on samples that were self-collected; In addition, RT-PCR test (performed prior enrollment) results were obtained.
Period: Overall Study
Arm/Group | BIOZEK COVID-19 Antigen Rapid Test
Started | 185
Completed | 185
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- BIOZEK COVID-19 Antigen Rapid Test (Oral Fluid): BIOZEK COVID-19 Antigen Rapid Test performed by subjects on self-collected, oral fluid samples compared to RT-PCR.
Arm/Group | BIOZEK COVID-19 Antigen Rapid Test (Oral Fluid)
Number analyzed (Participants) | 185
Age, Customized [Count of Participants; unit: Participants]
  18-24 years | 36
  25-64 years | 128
  65-87 years | 19
  Unknown | 2
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data was not captured for 3 participants.
  Participants
    number analyzed (Participants) | 182
    Female | 111
    Male | 71
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Arabic | 1
  Asian | 12
  Black | 51
  Caucasian | 74
  Hispanic/Latino | 31
  Indian | 1
  Native American | 1
  Pacific Islander | 4
  Unknown | 10
Region of Enrollment [Number; unit: participants]
  United States | 185

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity and Specificity of Biozek Covid-19 Antigen Rapid Test (Saliva)
Description: The Biozek Antigen Rapid Tests performed by subjects on the self-collected, oral fluid samples . Sensitivity was calculated using (TP/TP+FN)*100% formula.
  Specificity was calculated using (TN/TN+FP)*100% formula.
Time Frame: 6 months
Measure: Number; unit: percentage - Sensitivity and specificity
Arm/Group | BIOZEK COVID-19 Antigen Rapid Test (Oral Fluid)
Number analyzed (Participants) | 185
percentage - Sensitivity and specificity
  Sensitivity | 97.5
  Specifity | 100

2. Primary Outcome: Sensitivity and Specificity of Biozek Covid-19 Antigen Rapid Test (Nasopharyngeal Swab)
Description: The Biozek Antigen Rapid Tests performed by subjects on the self-collected, nasopharyngeal samples . Sensitivity was calculated using (TP/TP+FN)*100% formula.
  Specificity was calculated using (TN/TN+FP)*100% formula.
Time Frame: 6 months
Measure: Number; unit: percentage - Sensitivity and specificity
Groups:
- BIOZEK COVID-19 Antigen Rapid Test (Oral Fluid): The Biozek Antigen Rapid Tests performed by subjects on the self-collected, nasopharyngeal samples . Sensitivity was calculated using (TP/TP+FN)*100% formula.
  Specificity was calculated using (TN/TN+FP)*100% formula.
Arm/Group | BIOZEK COVID-19 Antigen Rapid Test (Oral Fluid)
Number analyzed (Participants) | 185
percentage - Sensitivity and specificity
  Sensitivity | 97.8
  Specificity | 100

ADVERSE EVENTS:
Time Frame: 1 visit - up to 2 hours
Arm/Group | BIOZEK COVID-19 Antigen Rapid Test (Oral Fluid)
All-Cause Mortality (participants affected / at risk) | 0/185
Serious Adverse Events (participants affected / at risk) | 0/185
Other Adverse Events (participants affected / at risk) | 0/185

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/79/NCT04926779/Prot_SAP_000.pdf